CLINICAL TRIAL: NCT07259746
Title: A Multi-Institutional Longitudinal Randomized Controlled Trial of Student Well-Being Using the Flourish App
Brief Title: Study of Student Flourishing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flourish Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Flourish2025
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: well-being; digital; positive psychology; students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flourish app condition (Experimental): Participants in this condition will gain access to the Flourish app and be instructed to use it at least twice a week for 6 weeks.
  Interventions: Behavioral: Digital toolkit
- Flourish app with buddies condition (Experimental): Participants in this condition will gain access to the Flourish app and be instructed to use it at least twice a week for 6 weeks. In addition, they will be instructed to invite a buddy (e.g., friend, family member) to join them on the app.
  Interventions: Behavioral: Digital toolkit
- MHA Resources (Active Comparator): Participants in this condition will continue to use existing school resources and will be provided with information directing them to external Mental Health America (MHA) resources. Participants in this arm do not receive access to the Flourish app.
  Interventions: Behavioral: Mental Health America Resources

INTERVENTIONS:
Behavioral: Digital toolkit — A mobile application providing a science-based digital toolkit and AI chatbot.
  Other Names: Flourish app
  Arms: Flourish app condition; Flourish app with buddies condition
Behavioral: Mental Health America Resources — Access to national mental health resources from Mental Health America, which can be found here: https://mhanational.org/resources/.
  Arms: MHA Resources

SUMMARY:
The goal of this study is to learn how a science-based mobile app, called Flourish, affects student well-being.

The main questions it aims to answer are:

1. Does receiving access to the Flourish app increase well-being (e.g., positive affect, loneliness, belonging) among students?
2. Does using the Flourish app in combination with a human buddy/friend lead to better outcomes than using the app alone?

Researchers will compare three different groups to see if and how the Flourish app works to improve student well-being:

1. Waitlist Control Group: Students continue with existing school resources.
2. Flourish App Group: Students use the Flourish app (a digital toolkit and AI chatbot) twice per week.
3. Flourish App + Buddy Group: Students use the Flourish app twice per week with someone else as a "Flourish Buddy".

Participants will:

Be randomly assigned to one of the three groups listed above. Use the app or continue with regular resources for 6 weeks. Complete four short online surveys about their well-being (at the beginning, during the 6 weeks, and at the end).

ELIGIBILITY:
Inclusion Criteria:

* Currently a student at one of the participating institutions
* Age 18 or older
* Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Subcomponents of Affect Scale | Baseline, bi-weekly for 6 weeks (3 time points)
  The Subcomponents of Affect Scale (SAS) is an 18-item measure of affect, divided into nine positive and nine negative adjectives. Positive subscales include calm, well-being, and vigor, while negative subscales include depression, anxiety, and anger. Participants rate each adjective from 0 (not at all accurate) to 4 (extremely accurate) based on their feelings over the past two weeks. Total scores for positive and negative affect are summed from their subscales.
Implicit Theories of Emotion | Baseline and 6 weeks post-baseline
  Implicit theories of emotion were assessed using the Implicit Theories of Emotion Scale, adapted from Dweck's Implicit Theories of Intelligence framework. The scale includes four items assessing beliefs about whether emotions are malleable (incremental) or fixed (entity). Participants rate each item on a 6-point scale from 1 ("Strongly disagree") to 6 ("Strongly agree"). The two entity items are reverse-scored, and all items are averaged to create a single score ranging from 1 to 6, with higher scores indicating stronger endorsement of an incremental (malleable) theory of emotion.
Loneliness | Baseline, bi-weekly for 6 weeks (3 time points)
  The UCLA 3-Item Loneliness Scale is a brief measure assessing subjective feelings of loneliness and social isolation. Participants rate each item on a 3-point scale, from 1 (hardly ever) to 3 (often), with higher scores indicating greater loneliness.
Perceived Cohesion | Baseline, 6 weeks post-baseline
  The Perceived Cohesion Scale measures a sense of belonging and morale within a community using a Likert scale from 0 (strongly disagree) to 10 (strongly agree). For our purposes, we use a single-item version: "I see myself as part of the campus community."
Closeness to University | Baseline and 6 weeks post-baseline
  Closeness to one's university was assessed using a modified single-item Inclusion of Other in the Self measure. Participants were shown seven pairs of increasingly overlapping circles and asked, "Which picture best describes your relationship with your university?" Responses range from 1 to 7, with higher scores indicating greater perceived closeness to the university.
Perceived Social Support (PSSS-3) | Baseline, bi-weekly for 6 weeks (3 time points)
  Perceived social support was assessed using a 3-item short form based on the ACO (PSSS-A6) and adapted from the Multidimensional Scale of Perceived Social Support (MSPSS). Participants rate each item on a 7-point scale from 1 ("Very Strongly Disagree") to 7 ("Very Strongly Agree"). Total scores are summed, yielding a range from 3 to 21, with higher scores indicating greater perceived social support.
Mindfulness (Mindful Attention Awareness Scale) | Baseline and 6 weeks post-baseline
  Mindfulness was assessed using a 5-item short form of the Mindful Attention Awareness Scale (MAAS), modified to assess experiences over the past two weeks. Participants rate each item on a 7-point scale from 0 ("Not at all") to 6 ("Very much"). Items are averaged to create a total score ranging from 0 to 6, with higher scores reflecting lower mindfulness. For interpretability in analyses, this score is reverse-scored so that higher values indicate greater mindfulness.
Resilience | Baseline, 6 weeks post-baseline
  The Brief Resilience Scale (BRS) is a 6-item measure of stress recovery, rated from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate a stronger ability to "bounce back" after setbacks.
Flourishing Scale | Baseline, 6 weeks post-baseline
  The Flourishing Scale is an 8-item measure of psychological well-being. Respondents rate items from 1 ("Strongly disagree") to 7 ("Strongly agree"), yielding a total score range from 8 to 56. Higher scores indicate greater well-being and flourishing.
Retention / Enrollment Intention | Baseline, 6 weeks post-baseline
  Retention intention was assessed using 2 items evaluating students' likelihood of continuing their enrollment. Participants respond to "How likely are you to stay enrolled next quarter/semester?" on a 5-point scale from 1 ("Very unlikely") to 5 ("Very likely"). A second item asks, "How often have you considered leaving your college/university in the past semester?" rated from 1 ("Never") to 5 ("Very often"). Higher scores on the first item indicate greater intention to persist, while higher scores on the second item indicate greater consideration of leaving.

SECONDARY OUTCOMES:
Depression (PHQ-2) | Baseline, bi-weekly for 6 weeks (3 time points)
  The PHQ-2 is an 2-item measure assessing depression severity over the past two weeks. Each item scores from 0 ("not at all") to 3 ("nearly every day"), with total scores from 0 to 6. Higher scores indicate greater depression severity.
Anxiety (GAD-2) | Baseline, bi-weekly for 6 weeks (3 time points)
  The GAD-2 (Generalized Anxiety Disorder-2) is a 2-item measure assessing anxiety severity. Each item is rated from 0 ("not at all") to 3 ("nearly every day"), with total scores ranging from 0 to 6. Higher scores indicate greater anxiety severity.
Perceived Stress (PSS-4) | Baseline, bi-weekly for 6 weeks (3 time points)
  The PSS-4 (Perceived Stress Scale-4) is a 4-item measure of perceived stress, rated from 0 ("never") to 4 ("very often"). Scores range from 0 to 16, with higher scores indicating greater stress.
Academic Self Efficacy | Baseline, 6 weeks post-baseline
  The 5-item Academic Self-Efficacy scale measures students' confidence in their ability to succeed academically. Participants rate their agreement with statements such as "I generally manage to solve difficult academic problems if I try hard enough" on a 5-point scale, from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater self-belief in tackling academic challenges and achieving study-related goals.
Satisfaction With Life | Baseline, bi-weekly for 6 weeks (3 time points)
  Life satisfaction was assessed using a single-item measure asking, "All things considered, how satisfied are you with your life as a whole?" Participants respond on an 11-point scale from 0 ("Completely dissatisfied") to 10 ("Completely satisfied"). Higher scores indicate greater overall life satisfaction.
School Perceptions | Baseline, 6 weeks post-baseline
  School perceptions are measured using two single-item measures from the Healthy Minds Survey. The first item rates satisfaction with the overall school experience from 1 (very dissatisfied) to 6 (very satisfied). The second item rates agreement with the statement, "At my school, students' mental and emotional well-being is a priority," on a scale from 1 (strongly agree) to 6 (strongly disagree).
Multi-Dimensional Measure of Trust | 6 weeks post-baseline
  The Multi-Dimensional Measure of Trust (MDMT) assesses perceived trustworthiness of the Flourish chatbot, Sunnie, through a set of 10 attributes (Form A), rated from 0 (Not at all) to 5 (Very), with a 'Does Not Fit' option. Only participants in the intervention conditions (Flourish app; Flourish app + buddies conditions) complete this measure.
Expectations and Experiences of Chatbots | Baseline, 6 weeks post-baseline
  This measure, adapted from the Working Alliance Inventory - Short Revised (WAI-SR), assesses participants' expectations and experiences with chatbots. Participants rate anticipated and actual interactions across three areas-Goal, Task, and Bond-on a 5-point scale from 1 (seldom) to 5 (always), with higher scores indicating stronger alignment.
Perceived Empathy of Sunnie | 6 weeks post-baseline
  Perceived empathy toward the Flourish chatbot, Sunnie, will be assessed using a 7-item measure. Participants rate each item from 1 ("Strongly disagree") to 6 ("Strongly agree"). Items are averaged to create a composite score, with higher scores indicating greater perceived empathy. This was only presented to those in the intervention conditions.
Flourish Buddy Responsiveness | Weeks 4 and 6 post-baseline
  For participants with at least one Flourish Buddy, responsiveness of the selected buddy will be assessed using a 3-item measure assessing how accepted, understood, and cared for participants feel by their buddy. Items are rated from 1 ("Not at all") to 7 ("Very much") and averaged; higher scores indicate greater perceived responsiveness.
Relationship Satisfaction with Flourish Buddy | Weeks 4 and 6 post-baseline
  For participants with at least one Flourish Buddy, relationship satisfaction with the selected buddy will be assessed using RAS-1, a single item rating overall satisfaction with the relationship from 1 ("Not satisfied") to 5 ("Very satisfied"). Higher scores indicate greater satisfaction.
Perceived Relationship Improvement | 6 weeks post-baseline
  Perceived improvement in the relationship with an existing Flourish Buddy will be assessed using a single item ("To what extent did being Flourish Buddies with this person improve your relationship?"). This item is shown to participants in either Flourish condition who reported having a Flourish Buddy. Participants rate the item from 1 ("Not at all") to 7 ("Very much"). Higher scores indicate greater perceived improvement.

OTHER OUTCOMES:
Net Promoter Score (NPS) | 6 weeks post-baseline
  Intervention satisfaction will be assessed using the Net Promoter Score (NPS). Participants in the intervention and control conditions will respond to the item: "How likely are you to recommend the Flourish app / MHA resources to a friend or colleague?" on an 11-point scale from 0 ("Not at all likely") to 10 ("Extremely likely"). Higher scores indicate greater likelihood of recommending the intervention.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - University of California, Berkeley, Berkeley, California
  - Foothill College, Los Altos Hills, California
  - Chapman University, Orange, California
  - University of Colorado Denver, Denver, Colorado
  - University of Hawai'i at Mānoa, Honolulu, Hawaii
  - Kansas State University, Manhattan, Kansas
  - Brown University, Providence, Rhode Island
  - University of Washington, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
- University of Victoria, Victoria, British Columbia, Canada
- University of Canterbury, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified participant data on OSF from each study timepoint across both conditions, including all data used in our analyses.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning upon submission for publication with no end date.